CLINICAL TRIAL: NCT00246493
Title: Vascular Aging: The Link That Bridges Age to Atherosclerosis (The VALIDATE Study)
Status: Terminated | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904294; 04-AG-N294
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2017-11-01

CONDITIONS: Atherosclerosis; Cardiovascular Disease; Vascular Diseases
Keywords: Coronary; Endothelial; Vascular; Atherosclerosis; Arterial
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The prevalence, incidence, and severity of atherosclerotic disease all markedly increase with age. Basic experimental and observational data demonstrate that aging magnifies the pathologic and clinical consequences of established risk factors and is the most potent individual risk factor for coronary atherosclerosis and for adverse outcomes following an ischemic event. These findings suggest that normal aging alters the vascular substrate so as to promote the development and progression of atherosclerosis. The age-associated changes in vascular structure and function include an increase in central vascular stiffness, intimal proliferation, and endothelial dysfunction. The major hypothesis is that the above alterations in vascular substrate (i.e. vascular age) are an important determinant of the age associated increased likelihood for the development and progression of coronary atherosclerotic disease.

This program will non-invasively characterize vascular age and atherosclerotic burden in BLSA participants and individuals with successful aging, i.e. those with no or minimal evidence of coronary atherosclerotic disease, and those with premature, clinically evident coronary artery disease. It will repeat measures of vascular age and atherosclerotic burden three years after the first assessment. By examining the impact of vascular age on the initial extent and the progression of atherosclerotic burden over a two to three-year period, it will test the hypothesis that vascular age is an important determinant of the ageassociated increase in atherosclerotic disease....

DETAILED DESCRIPTION:
The prevalence, incidence, and severity of atherosclerotic disease all markedly increase with age. Basic experimental and observational data demonstrate that aging magnifies the pathologic and clinical consequences of established risk factors and is the most potent individual risk factor for coronary atherosclerosis and for adverse outcomes following an ischemic event. These findings suggest that normal aging alters the vascular substrate so as to promote the development and progression of atherosclerosis. The age-associated changes in vascular structure and function include an increase in central vascular stiffness, intimal proliferation, and endothelial dysfunction. The major hypothesis is that the above alterations in vascular substrate (i.e. vascular age) are an important determinant of the age associated increased likelihood for the development and progression of coronary atherosclerotic disease.

This protocol will non-invasively characterize vascular age and atherosclerotic burden in BLSA participants and individuals with successful aging, i.e. those with no or minimal evidence of coronary atherosclerotic disease, and those with premature, clinically evident coronary artery disease. It will repeat measures of vascular age and atherosclerotic burden three years after the first assessment. By examining the impact of vascular age on the initial extent and the progression of atherosclerotic burden over a two to three-year period, it will test the hypothesis that vascular age is an important determinant of the age-associated increase in atherosclerotic disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

For all groups:

1. Age 30 years or older
2. Ability and willingness to participate in the protocol and undergo vascular studies and chest MDCT examinations

For the second group:

1) Coronary artery calcium score of zero or less than 25th percentile of that expected based on age and gender.

For the third group:

1) Coronary artery calcium score which is greater than the 50th percentile of that computed based on age and gender, or known coronary disease on the basis of:

i. prior documented myocardial infarction or

ii. typical ischemic symptoms and catheterization documented stenosis of greater than or equal to 70% in at least one major coronary artery

If male, diagnosis was made under 50 years of age

If female, diagnosis was made under 60 years of age.

EXCLUSION CRITERIA

1. Atrial fibrillation (due to limitations with gating on MDCT)
2. For the first 2 groups: History of procedures used for treatment of CVD (CABG, angioplasty, pacemaker or defibrillator implantation, any surgery on the heart or the arteries)
3. Active treatment for cancer
4. Serious medical condition which could hinder participation or make it unlikely that they will live for three years (for f/u)
5. Weight>300 lb (maximum weight allowed on CT tables)
6. Inability to provide an informed consent
7. For females, current pregnancy because of the radiation associated with the helical CT and the unknown risks to a fetus. This is only temporary, and women wishing to participate may be enrolled six weeks after delivery.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2004-06-22; Study Completion 2017-11-01

PRIMARY OUTCOMES:
Characterize vascular age relat-BLSA | Two-three years

SECONDARY OUTCOMES:
Characterize vascular age relat-other | Two-three years

CONTACTS AND LOCATIONS:
Overall Officials: Edward G Lakatta, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - National Institute of Aging, Clinical Research Unit, Baltimore, Maryland

REFERENCES:
- [Background] Lakatta EG. Cardiovascular aging research: the next horizons. J Am Geriatr Soc. 1999 May;47(5):613-25. doi: 10.1111/j.1532-5415.1999.tb02579.x. No abstract available. PMID 10323658
- [Background] Franklin SS, Wong ND, Larson MG, Kannel WB, Levy D. How important is pulse pressure as a predictor of cardiovascular risk? Hypertension. 2002 Feb;39(2):E12-3. No abstract available. PMID 11847204
- [Background] Grundy SM. Coronary plaque as a replacement for age as a risk factor in global risk assessment. Am J Cardiol. 2001 Jul 19;88(2A):8E-11E. doi: 10.1016/s0002-9149(01)01712-x. PMID 11473737